CLINICAL TRIAL: NCT06834191
Title: Analysis of the Relationship Between Immunosuppressive Treatment Status and Clinical Course of Parkinson's Disease
Brief Title: Relationship Between Immunosuppressive Treatment Status and Clinical Course of Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/164/2024
Record Dates: First submitted 2025-01-31; First posted 2025-02-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-01

CONDITIONS: Parkinson Disease
Keywords: Immunosuppression; Immunosuppressive treatment; cross-sectional study; observational study; Parkinson disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Parkinson's receiving long - term immunosuppressive treatment - study group
- People with Parkinson's without long-term immunosuppressive treatment history - control group

SUMMARY:
The goal of this observational study is to learn if immunosuppressive drug treatment influences the clinical course of Parkinson's disease. Recent research suggests that Parkinson's disease may have an inflammatory background. Numerous studies have identified elevated levels of pro-inflammatory markers in people with Parkinson's disease. Therefore, immunosuppressive drugs may potentially affect the course of this disease.

The investigators will recruit people with Parkinson's disease, who receive long-term immunosuppressive treatment for other chronic illnesses, into the study group. The study will also recruit people with Parkinson's disease with no history of immunosuppressive drug treatment into the control group. The main question this study aims to answer is:

> Does immunosuppressive drug treatment slow down the onset and/or progression of Parkinson's disease?

Researchers will compare Parkinson's disease progression rates and serum inflammatory marker levels between the study and control group, to see if immunosuppressive drug treatment influences the course of Parkinson's disease.

The study requires each participant to attend one hospital appointment. This appointment will be approximately one hour long, and will involve:

1. clinical Parkinson's disease motor assessments conducted by the research team -> participants will be evaluated in the OFF state, meaning they will not have taken their Parkinson's disease medication the day of the assessment;
2. completion of Parkinson's disease symptom scales;
3. a one-time serum sample collection;
4. detailed medical history obtainment from the participant by the research team, with a primary focus on the patient's immunosuppressive treatment history and individual clinical course of Parkinson's disease.

ELIGIBILITY:
Inclusion criteria for the study group:

1. Diagnosis of Parkinson's disease according to the International Parkinson and Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's disease;
2. Immunosuppressive medication use - medication taken regularly, which we have defined as administered at a dose and frequency effective for the indicated disease, for over 12 months, systemic administration route (oral, intramuscular, subcutaneous, intravenous and inhaled); The most commonly used immunosuppressive drugs that we anticipate will be used by the study group participants include: glucocorticosteroids (GC) - budesonide, cortisone, dexamethasone, hydrocortisone, methylprednisolone, prednisolone, prednisone, triamcinolone; calcineurin inhibitors - tacrolimus, cyclosporine; inosine monophosphate dehydrogenase (IMDH) inhibitors - azathioprine, leflunomide, mycophenolate; mammalian target of rapamycin (mTOR) inhibitors - sirolimus, everolimus; biologics - abatacept, adalimumab, anakinra, certolizumab, etanercept, infliximab, ixekizumab, natalizumab, rituximab, secukinumab, tocilizumab, ustekinumab, vedolizumab; antimetabolites - methotrexate; inclusion of participants taking immunosuppressive drugs not listed above will be considered individually;
3. Provision of informed consent to participate in the study.

Inclusion criteria for the control group:

1. Diagnosis of Parkinson's disease according to the International Parkinson and Movement Disorder Society Clinical Diagnostic Criteria for Parkinson's Disease;
2. No history of regular use of immunosuppressive medications;
3. Provision of informed consent to participate in the study.

Exclusion criteria for the study group:

1. Immunosuppressive drug administration at an ad hoc basis (i.e. when symptoms occur) or irregularly (i.e. drug taken at an inappropriate dose and/or with a regularity ineffective for the indicated disease);
2. Use of immunosuppressive drugs for a period of less than 12 months;
3. Ineffective treatment of the disease requiring the use of immunosuppressive drugs (no improvement/progression of disease symptoms);

Additional exclusion criteria for both the study and control groups:

1. Advanced cancer; severe heart failure; severe renal failure; untreated autoimmune disease; active inflammation; diseases that impair drug absorption/metabolism;
2. Dementia;
3. Failure/inability to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited among patients of the Department of Neurology and Parkinsonism Clinic of the Faculty of Health Sciences, Medical University of Warsaw, Warsaw, Poland
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Annual motor progression rate - Unified Parkinson's Disease Rating Scale PART III OFF | Day 1
  This primary outcome will measure annual Parkinson's disease motor symptom progression rates using Part III (Motor Examination) of the Unified Parkinson's Disease Rating Scale (UPDRS). Assessments will be conducted in the OFF state, meaning the participant will not have taken any Parkinson's disease medication the day of the assessment. Part III of the UPDRS contains 18 items, the minimum value of UPDRS Part III is 0 points, and the maximum value is 132 points. In UPDRS Part III the higher the score, the worse the outcome. Annual progression rates will be calculated based on the time from the participant's motor symptom onset to the time of the appointment.
Annual LEDD increase rate | Day 1
  This secondary outcome will measure annual Parkinson's disease levodopa equivalent daily dose (LEDD) increase rates for each participant. Parkinson's disease medication taken by the participant will be procured at each participant's individual appointment. LEDD values will then be calculated based on the doses and types of Parkinson's disease medication taken by the participant. Annual LEDD rates will be calculated based on the LEDD value and time from the participant's motor symptom onset to the time of the appointment.
Age of motor symptom onset | Day 1
  This secondary outcome will measure the age of onset of Parkinson's disease motor symptoms.

SECONDARY OUTCOMES:
Annual motor progression rate - Hoehn and Yahr scale | Day 1
  This primary outcome will measure annual Parkinson's disease motor symptom progression rates using the Hoehn and Yahr scale. This scale is used for staging functional disability associated with Parkinson's disease. The stages range from 1 to 5, and the higher the score the worse the outcome. Annual progression rates will be calculated based on the time from the participant's motor symptom onset to the time of the appointment.
Annual motor progression rate - Unified Parkinson's Disease Rating Scale PART II | Day 1
  This primary outcome will measure annual Parkinson's disease motor symptom progression rates using Part II (Motor Aspects of Experiences of Daily Living ) of the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS). Part II of the MDS-UPDRS contains 13 items, the minimum value of MDS-UPDRS Part II is 0 points, and the maximum value is 52 points. In UPDRS Part II the higher the score, the worse the outcome. Annual progression rates will be calculated based on the time from the participant's motor symptom onset to the time of the appointment.
Serum inflammatory marker levels - IL-1β | Day 1
  This secondary outcome measures the level of IL-1β in each participant at a single time-point.
Serum inflammatory marker levels - IL-6 | Day 1
  This secondary outcome measures the level of IL-6 in each participant at a single time-point.
Serum inflammatory marker levels - calprotectin | Day 1
  This secondary outcome measures the level of calprotectin in each participant at a single time-point.
Serum inflammatory marker levels - TNFα | Day 1
  This secondary outcome measures the level of TNFα in each participant at a single time-point.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Faculty of Health Science, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brumm MC, Siderowf A, Simuni T, Burghardt E, Choi SH, Caspell-Garcia C, Chahine LM, Mollenhauer B, Foroud T, Galasko D, Merchant K, Arnedo V, Hutten SJ, O'Grady AN, Poston KL, Tanner CM, Weintraub D, Kieburtz K, Marek K, Coffey CS; Parkinson's Progression Markers Initiative. Parkinson's Progression Markers Initiative: A Milestone-Based Strategy to Monitor Parkinson's Disease Progression. J Parkinsons Dis. 2023;13(6):899-916. doi: 10.3233/JPD-223433. PMID 37458046
- [Background] Postuma RB, Berg D, Stern M, Poewe W, Olanow CW, Oertel W, Obeso J, Marek K, Litvan I, Lang AE, Halliday G, Goetz CG, Gasser T, Dubois B, Chan P, Bloem BR, Adler CH, Deuschl G. MDS clinical diagnostic criteria for Parkinson's disease. Mov Disord. 2015 Oct;30(12):1591-601. doi: 10.1002/mds.26424. PMID 26474316
- [Background] Dulski J, Heckman MG, Nowak JM, Wszolek ZK. Protective Effect of Glucocorticoids against Symptomatic Disease in CSF1R Variant Carriers. Mov Disord. 2023 Aug;38(8):1545-1549. doi: 10.1002/mds.29504. Epub 2023 Jun 13. PMID 37309919
- [Background] Racette BA, Gross A, Vouri SM, Camacho-Soto A, Willis AW, Searles Nielsen S. Immunosuppressants and risk of Parkinson disease. Ann Clin Transl Neurol. 2018 May 31;5(7):870-875. doi: 10.1002/acn3.580. eCollection 2018 Jul. PMID 30009205
- [Background] Bruggeman A, Vandendriessche C, Hamerlinck H, De Looze D, Tate DJ, Vuylsteke M, De Commer L, Devolder L, Raes J, Verhasselt B, Laukens D, Vandenbroucke RE, Santens P. Safety and efficacy of faecal microbiota transplantation in patients with mild to moderate Parkinson's disease (GUT-PARFECT): a double-blind, placebo-controlled, randomised, phase 2 trial. EClinicalMedicine. 2024 Mar 27;71:102563. doi: 10.1016/j.eclinm.2024.102563. eCollection 2024 May. PMID 38686220
- [Background] Schwiertz A, Spiegel J, Dillmann U, Grundmann D, Burmann J, Fassbender K, Schafer KH, Unger MM. Fecal markers of intestinal inflammation and intestinal permeability are elevated in Parkinson's disease. Parkinsonism Relat Disord. 2018 May;50:104-107. doi: 10.1016/j.parkreldis.2018.02.022. Epub 2018 Feb 12. PMID 29454662
- [Background] Franceschi C, Valensin S, Fagnoni F, Barbi C, Bonafe M. Biomarkers of immunosenescence within an evolutionary perspective: the challenge of heterogeneity and the role of antigenic load. Exp Gerontol. 1999 Dec;34(8):911-21. doi: 10.1016/s0531-5565(99)00068-6. PMID 10673145
- [Background] Qin XY, Zhang SP, Cao C, Loh YP, Cheng Y. Aberrations in Peripheral Inflammatory Cytokine Levels in Parkinson Disease: A Systematic Review and Meta-analysis. JAMA Neurol. 2016 Nov 1;73(11):1316-1324. doi: 10.1001/jamaneurol.2016.2742. PMID 27668667
- [Background] Brodacki B, Staszewski J, Toczylowska B, Kozlowska E, Drela N, Chalimoniuk M, Stepien A. Serum interleukin (IL-2, IL-10, IL-6, IL-4), TNFalpha, and INFgamma concentrations are elevated in patients with atypical and idiopathic parkinsonism. Neurosci Lett. 2008 Aug 22;441(2):158-62. doi: 10.1016/j.neulet.2008.06.040. Epub 2008 Jun 19. PMID 18582534
- [Background] Tansey MG, Wallings RL, Houser MC, Herrick MK, Keating CE, Joers V. Inflammation and immune dysfunction in Parkinson disease. Nat Rev Immunol. 2022 Nov;22(11):657-673. doi: 10.1038/s41577-022-00684-6. Epub 2022 Mar 4. PMID 35246670